CLINICAL TRIAL: NCT04481815
Title: Efficacy and Safety Study of Lenalidomide Plus Rituximab and Methotrexate Chemotherapy（R2-MTX） Versus Rituximab and Methotrexate Chemotherapy（R-MTX） in Newly Diagnosed Primary Central Nervous System Lymphoma: a Multicenter, Open-Label, Randomised Phase 2 Study
Brief Title: Rituximab Plus Methotrexate With or Without Lenalidomide in Treating Patients With Newly Diagnosed Primary Central Nervous System Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IR2020001238
Record Dates: First submitted 2020-07-13; First posted 2020-07-22 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-10

CONDITIONS: PCNSL
Keywords: PCNSL; Lenalidomide
MeSH Terms: interventions — Rituximab; Lenalidomide; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- R2-MTX (Experimental): Experimental arm will be treated with R2-MTX regimen(Lenalidomide plus Rituximab and Methotrexate) for 6 cycles as initiate induction.If the patients achieved complete remission（CR）or partial remission（PR）with additional whole-brain radiotherapy（WBRT）, they processed to R2 maintenance(Lenalidomide plus Rituximab) for 4 cycles.
  Interventions: Drug: Rituximab; Drug: Lenalidomide; Drug: Methotrexate
- R-MTX (Sham Comparator): Control arm will be treated with R-MTX regimen(Rituximab and Methotrexate) for 6 cycles as initiate induction.If the patients achieved CR or PR with additional WBRT, they processed to Lenalidomide maintenance for 4 cycles.
  Interventions: Drug: Rituximab; Drug: Methotrexate

INTERVENTIONS:
Drug: Rituximab — 375mg/m2 intravenous infusion d1, every 3 weeks for 1 cycle, 6 cycles will be prescribed for induction therapy. 375mg/m2 intravenous infusion d1, every 8 weeks for 1 cycle, 4 cycles will be prescribed for maintenance therapy.
Drug: Lenalidomide — 25mg orally d1-10 every 3 weeks for 1 cycle, 6 cycles will be prescribed for induction therapy. 25mg orally d1-14,d29-42 every 8 weeks for 1 cycle, 4 cycles will be prescribed for maintenance therapy.
  Arms: R2-MTX
Drug: Methotrexate — 3.5g/m2 intravenous infusion for 4 hours in d1, every 21 days for 1 cycle, 6 cycles will be prescribed.

SUMMARY:
It is a multicenter, open-Label, randomised phase 2 study to compare the efficacy and safety study of R2-MTX chemotherapy（Lenalidomide, Rituximab and Methotrexate）with R-MTX chemotherapy（Rituximab and Methotrexate ）as first-line regimens in the treatment of newly diagnosed primary central nervous system lymphoma.2-year Progression free survival (PFS) is the primary endpoint.

DETAILED DESCRIPTION:
This is a multicenter, open-Label, randomised phase 2 study designed to evaluate the efficacy and safety of rituximab plus methotrexate with or without lenalidomide as first-line regimens in the treatment of primary central nervous system lymphoma. A total of 240 patients plan to participate in this study to receive a total 6 cycles of induction chemotherapy followed by 4 cycles of maintenance chemotherapy. Follow-ups should be taken up to the first 3 years.The primary endpoints were 2-year PFS rate and and secondary endpoints including objective response rate (ORR), PFS, overall survival (OS), and adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed Primary Central Nervous System (CNS) lymphoma
2. Age range 18-75 years old.
3. Eastern Cooperative Oncology Group performance status 0 to 3.
4. Previously untreated. Patients treated with steroid alone are eligible.
5. Patient's who are not planned to undergo consolidation with autologous hematopoietic stem cell transplantation（HSCT）.
6. Measurable disease was defined as at least ≥1.0cm in short-diameter by MRI.
7. Life expectancy of ≥ 3 months (in the opinion of the investigator).
8. Participants must be able to understand and be willing to sign a written informed consent document.
9. Women of reproductive potential must agree to use highly effective methods of birth control during the period of therapy and for 6 months after the last dose of the study drug. Men who are sexually active must agree to use highly effective contraception during the period of therapy and for 6 months after the last dose.
10. Women of childbearing potential must have a negative plasma pregnancy test upon study entry.
11. Adequate renal function: Estimated glomerular filtration rate (GFR) or estimated creatinine clearance (CrCl) ≥ 50 mL/min;Serum creatinine ≤ 2 times the upper limit of normal.
12. Adequate liver functions: Transaminase (AST/ALT) < 3 X upper normal value & Bilirubin < 2 X upper normal value.
13. Adequate hematological function: hemoglobin ≥ 9 g/dL absolute neutrophil count (ANC) ≥ 1,500/μL and platelet count ≥ 75,000/μL.

Exclusion Criteria:

1. Patient with systemic, non-CNS lymphoma metastatic to the CNS.
2. Patient is concurrently using other approved or investigational antineoplastic agents.
3. Presence of active hepatitis B virus(HBV) infection (HBsAg positive and HBV-DNA≥ 104), hepatitis C virus(HCV) infection, acquired and congenital immunodeficiency diseases include but not limited to HIV.
4. Patient is allergic to components of the study drug.
5. Patient has an active concurrent malignancy requiring active therapy.
6. Patient has significant abnormalities on screening electrocardiogram (EKG) and active and significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, uncontrolled congestive heart failure, uncontrolled hypertension, valvular disease, pericarditis, or myocardial infarction within 6 months of screening.
7. Patient is known to have an uncontrolled active systemic infection.
8. Patient has a life-threatening illness, medical condition, or organ system dysfunction that, in the opinion of the investigator, could compromise the subject's safety or put the study outcomes at undue risk.
9. Women who are pregnant or nursing (lactating), where pregnancy is defined as a state of a female after conception until the termination of gestation, confirmed by a positive plasma human chorionic gonadotropin(hCG) laboratory test of > 5 mIU/mL.
10. The patient is unwell or unable to participate in all required study evaluations and procedures.
11. Drug abuse, medical, psychological or social conditions which may interfering with subjects' participation in the study or evaluation of the results.
12. Patients considered unsuitable to participate in the study by the researchers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
2-year progression free survival | 2 years
  From date of patients sign informed consent until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years

SECONDARY OUTCOMES:
Objective response rate | At the end of Cycle 6 chemotheray
  At the end of Cycle 6 (each cycle is 21 days) the ratio of numbers of patients with complete response and partial response to all the participants receiving treatment
Overall survival | 3 years
  From date of patients sign informed consent until the date of death or the date of last follow-up time, whichever came first, assessed up to 3 years
Progression free survival | 3 years
  From date of patients sign informed consent until the date of progression or death or the date of last follow-up time, whichever came first, assessed up to 3 years
Treatment-related adverse events | 1 year
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

OTHER OUTCOMES:
Serum ctDNA biomarkers and tissue biomarkers | Up to 3 years
  Next generation sequencing of serum and tissue samples to identify circulating tumor DNA（ctDNA）and tissue biomarkers before and after treatment

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No